CLINICAL TRIAL: NCT02862522
Title: Clinical Follow-up of Patients With Assessment of Endothelial Dysfunction/Coronary Spasm
Brief Title: Uric Acid Levels and Endothelial Functions
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amir Lerman, Professor of Medicine, Mayo Clinic
Other Study IDs: 05-004191; R01HL092954 (NIH); R01AG031750 (NIH)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
Keywords: uric acid; microvascular dysfunction; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women With CED: All subjects had blood work with included measurement of C-reactive protein, complete blood count with differential, basic chemistry panel, and uric acid level. All subjects completed a standardized questionnaire to assess baseline characteristics. All subjects underwent comprehensive coronary endothelial function assessment. Subjects completed a questionnaire of overall health several years after the index coronary angiogram and endothelial function study.
  Interventions: Other: Questionnaire of overall health
- Women Without CED: All subjects had blood work with included measurement of C-reactive protein, complete blood count with differential, basic chemistry panel, and uric acid level. All subjects completed a standardized questionnaire to assess baseline characteristics. All subjects underwent comprehensive coronary endothelial function assessment. Subjects completed a questionnaire of overall health several years after the index coronary angiogram and endothelial function study.
  Interventions: Other: Questionnaire of overall health

INTERVENTIONS:
Other: Questionnaire of overall health — The standardized questionnaire was used to assess occurrence of major adverse cardiovascular events including stroke, re-hospitalization, myocardial infarction or death. Responses were verified by medical record review conducted by an investigator blinded to the results of the standardized questionnaire.

SUMMARY:
Uric acid is a risk factor for coronary artery disease (CED) in postmenopausal women but the association with inflammation and coronary microvascular endothelial dysfunction is not well-defined. The aim of this study was to determine the relationship of serum uric acid, inflammatory markers and CED.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Mayo Clinic for cardiac catheterization
* Postmenopausal

Exclusion Criteria:

* History of percutaneous coronary intervention
* Coronary artery bypass graft surgery
* Unstable angina pectoris
* Valvular heart disease
* Peripheral vascular disease
* Known congestive heart failure

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients referred to Mayo Clinic's cardiac care clinic in Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 1992-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Serum Uric Acid Level | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided